CLINICAL TRIAL: NCT04035135
Title: A Phase 1b Study to Evaluate the Safety, Tolerability and Drug-Drug Interactions of ANX005 and Intravenous Immunoglobulin (IVIg) in Subjects With Guillain Barré Syndrome
Brief Title: A Clinical Study of ANX005 and IVIG in Subjects With Guillain Barré Syndrome (GBS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Annexon, Inc. (Industry)
Collaborators: ResearchPoint Global (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANX005-GBS-03
Record Dates: First submitted 2019-07-11; First posted 2019-07-29 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Guillain-Barré Syndrome
MeSH Terms: conditions — Guillain-Barre Syndrome | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Intervention Model Description: Open label combination treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label Treatment Arm (Experimental): One (1) dose of ANX005, 75 mg/kg, will be administered IV. IVIg, 0.4 g/kg, will be administered for 5 consecutive Days.
  Interventions: Drug: ANX005; Drug: Intravenous immunoglobulin

INTERVENTIONS:
Drug: ANX005 — investigational drug
  Other Names: Anti C1q Antibody
Drug: Intravenous immunoglobulin — investigational drug
  Other Names: IVIg

SUMMARY:
This study is a multi center, open-label, study of ANX005 in combination with IVIg in subjects diagnosed with GBS.

DETAILED DESCRIPTION:
The study will enroll approximately 12 subjects into one cohort, with subjects receiving 75 mg/kg of ANX005, a dose shown to be safe and well-tolerated as monotherapy and that provides a meaningful level of exposure to be tested in combination with IVIg. Dosing of IVIg will be administered as is the current standard of care (0.4 g/kg/day x 5 days) and ANX005 will be administered concurrently, beginning on Day 1 or 2 of the treatment period. Subjects will be followed for 6 months after treatment for observation and evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GBS according to the National Institute of Neurological Disorders and Stroke Diagnostic Criteria for Guillain Barré Syndrome
* Onset of GBS-related weakness ≤14 days prior to infusion
* GBS-DS score of 3, 4, or 5

Exclusion Criteria:

* Clinically significant findings that may interfere with the conduct of the study or the interpretation of the data
* Be at risk of suicide or self-harm
* Received previous treatment with plasma exchange for GBS
* Any diagnosis of a variant of GBS
* Have a history of anaphylaxis or severe systemic response to immunoglobulin
* Documented, clinically significant, pre-existing polyneuropathy from another cause
* Clinically significant intercurrent illness, medical condition, or medical history
* History of chronic use of steroid or immunosuppressant medication
* Active alcohol, drug, or substance abuse
* Females who are pregnant, breast feeding, or unable or unwilling to use highly effective methods of contraception throughout the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ANX005 when administered in combination with IVIg: incidence of TEAEs, SAEs, AE's | 6 months
  As measured by incidence of TEAEs, SAEs, AE's related to ANX005, SAE's related to ANX005, Grade 3 or higher AEs, Grade 3 or higher AEs related to ANX005, AEs leading to study or treatment discontinuation.

SECONDARY OUTCOMES:
Pharmacokinetics of ANX005 when administered in combination with IVIg | 3 months
  As measured by ANX005 serum concentrations
Pharmacodynamics of ANX005 when administered in combination with IVIg | 4 months
  As measured by CH50 and C1q serum concentrations
Values and change from baseline in Guillain-Barré Syndrome Disability Score (GBS-DS) by visit | 6 months
  The 6-point Guillain-Barré Syndrme Disability Score (GBS-DS) is a widely accepted and easily obtainable scoring system used to assess functional status of GBS subjects. The score is as follows: 0 = Healthy, 1 = Minor symptoms and capable of running, 2 = Able to walk independently 10 meters or more but unable to run, 3=Able to walk more than 10 meters across an open space with help, 4 = Bedridden or chair bound, 5 = Needing mechanical ventilation, 6 = death

CONTACTS AND LOCATIONS:
Overall Officials: Henk-André Kroon, MD, MBA, Study Director — Annexon, Inc.
Locations (2):
- National Institute of Neurosciences and Hospital, Dhaka, Bangladesh
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No